CLINICAL TRIAL: NCT00086749
Title: A Prospective Study Of The Effect Of Tamoxifen On Breast Density In Premenopausal Women
Brief Title: Effect of Tamoxifen on Breast Density in Premenopausal Women With Breast Cancer or High Risk for Breast Cancer
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Seema Khan, MD, Northwestern University
Other Study IDs: NCI 00B2; NU-NCI-00B2; NCI-00B2
Record Dates: First submitted 2004-07-08; First posted 2004-07-12 (Estimated); Last update posted 2012-07-11 (Estimated); Status verified 2012-07

CONDITIONS: Breast Cancer
Keywords: breast cancer; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Tamoxifen group

SUMMARY:
RATIONALE: High estrogen levels may be associated with dense breast tissue and an increased risk of developing breast cancer. Tamoxifen may be effective in reducing breast density by decreasing estrogen levels.

PURPOSE: This phase I trial is studying how well tamoxifen works in reducing breast density in premenopausal women with breast cancer or at high risk of developing breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine whether breast density, as measured by digital mammography, decreases in premenopausal women receiving tamoxifen for breast cancer or for breast cancer risk reduction.
* Determine whether breast density, as determined by a trained mammographer, decreases in patients treated with this drug.
* Correlate tamoxifen-induced symptoms in estrogen target tissue with change in salivary steroids in patients treated with this drug.

Secondary

* Determine the effect of this drug on salivary steroids in regularly cycling and amenorrheic patients.
* Correlate changes in breast density with tamoxifen-induced alterations in sex steroid levels, as measured in the saliva, of patients treated with this drug.

OUTLINE: Patients receive oral tamoxifen once daily. Treatment continues for 5 years in the absence of disease metastasis (patients with known breast cancer) or a diagnosis of breast cancer (patients undergoing risk reduction).

Patients undergo mammography to determine breast density at baseline, at 6 and 12 months, and then annually for 4 years. Patients also collect daily salivary samples during the 30-day periods surrounding the imaging studies to measure salivary estradiol and progesterone levels. The results of the salivary hormone studies are correlated with density changes at study completion.

PROJECTED ACCRUAL: A total of 100 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Initiating tamoxifen as the sole systemic treatment for breast cancer OR for breast cancer risk reduction
* Undergoing mammography at least annually
* No bilateral breast cancer or stage IV breast cancer
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 20 to 45

Sex

* Female

Menopausal status

* Premenopausal

  * No change in menstrual patterns within the past 6 months

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* Not pregnant or nursing

  * No planned pregnancy within the next 5 years
* No medical or psychiatric disorder that would preclude giving informed consent

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy for breast cancer

Endocrine therapy

* See Disease Characteristics
* No prior tamoxifen for more than 1 month in duration

Radiotherapy

* Not specified

Surgery

* Not specified

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women who are initiating tamoxifen on the advice of their treating physician as the sole systemic treatment for breast carcinoma or breast cancer risk reduction
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2003-02; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Seema A. Khan, MD, Principal Investigator — Robert H. Lurie Cancer Center
Locations (1):
- Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois, United States